CLINICAL TRIAL: NCT00342407
Title: The Incidence of Breast and Other Cancers Among Female Flight Attendants
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902039; 02-C-N039
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Thyroid Cancer; Breast Cancer; Non-Melanoma Skin Cancer; Melanoma
Keywords: Cancer Risk; Cosmic Radiation; Airlines; Flight Attendants; Circadian Rhythm
MeSH Terms: conditions — Thyroid Neoplasms; Breast Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

GROUPS / COHORTS (1):
- Cohort: Female flight attendants

SUMMARY:
Flight attendants may be at an increased risk of breast and other cancers due to work-place exposures including cosmic radiation and circadian rhythm disruption form traveling across multiple time zones. This cancer incidence study will determine whether female flight attendants are at increased risk of breast and other cancers and whether the risk is dose-related. The study will include a cohort of approximately 10,000 women who were employed as flight attendants for one or more years.

Breast cancer cases will be identified from telephone interviews of living subjects and next-of-kin of deceased subjects, as well as from death certificates. The interview will also provide information about non-occupational risk factors for breast cancer such as parity. Both internal and external comparisons will be made. The primary analysis will evaluate the risk associated with occupational exposure within the cohort, controlling for non-occupational risk factors by stratification or modeling. The secondary analysis will compare the incidence of breast cancer in the cohort to that in the general population, with adjustment for factors such as lower parity which might increase breast cancer risk in the cohort independent of occupational exposure to cosmic radiation and circadian rhythm disruption. The risk of other ionizing radiation-related cancers, such as leukemia, lung cancer, and thyroid cancer, among flight attendants will also be evaluated. The results of the study will apply to female flight crew and frequent fliers.

DETAILED DESCRIPTION:
Flight attendants may be at an increased risk of breast and other cancers due to work-place exposures including cosmic radiation and circadian rhythm disruption from traveling across multiple time zones. This cancer incidence study will determine whether female flight attendants are at increased risk of breast and other cancers and whether the risk is dose-related. The study will include a cohort of approximately 9,631 women who were employed as flight attendants for one or more years.

Breast cancer cases will be identified from telephone interviews of living subjects and next-of-kin of deceased subjects, as well as from death certificates. The interview will also provide information about non-occupational risk factors for breast cancer such as parity. Both internal and external comparisons will be made. The primary analysis will evaluate the risk associated with occupational exposure within the cohort, controlling for non-occupational risk factors by stratification or modeling. The secondary analysis will compare the incidence of breast cancer in the cohort to that in the general population, with adjustment for factors such as lower parity which might increase breast cancer risk in the cohort independent of occupational exposure to cosmic radiation and circadian rhythm disruption. The risk of other ionizing radiation-related cancers, such as leukemia, lung cancer, and thyroid cancer, among flight attendants will also be evaluated. The results of the study will apply to female flight crew and frequent fliers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Employed as a flight attendant for one or more years by Pan AM before Pan Am ceased operation in 1991. For flight attendants who transferred to Pan Am from National Airlines when Pan Am bought National Airlines in 1981, the time employed as a flight attendant at National Airlines will be counted towards the one year minimum.

A U.S. citizen when they began working at Pan Am (or National Airlines, if the flight attendant transferred to Pan AM from National Airlines).

Worked at least one day after January 1, 1953.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female flight attendants
Sampling Method: Probability Sample
Enrollment: 6093 (Actual)
Dates: Start 2001-11-06 (Actual); Primary Completion 2005-12-31 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Breast and other cancers | Time of questionnaire, time of death
  survival

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Little, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institute for Occupational Safety and Health (NIOSH), Cincinnati, Ohio, United States

REFERENCES:
- [Background] Grajewski B, Waters MA, Whelan EA, Bloom TF. Radiation dose estimation for epidemiologic studies of flight attendants. Am J Ind Med. 2002 Jan;41(1):27-37. doi: 10.1002/ajim.10018. PMID 11757053
- [Background] Pinkerton LE, Waters MA, Hein MJ, Zivkovich Z, Schubauer-Berigan MK, Grajewski B. Cause-specific mortality among a cohort of U.S. flight attendants. Am J Ind Med. 2012 Jan;55(1):25-36. doi: 10.1002/ajim.21011. Epub 2011 Oct 10. PMID 21987391
- [Background] Waters MA, Grajewski B, Pinkerton LE, Hein MJ, Zivkovich Z. Development of historical exposure estimates of cosmic radiation and circadian rhythm disruption for cohort studies of Pan Am flight attendants. Am J Ind Med. 2009 Oct;52(10):751-61. doi: 10.1002/ajim.20738. PMID 19722196